CLINICAL TRIAL: NCT04861610
Title: Mindfulness-Based Intervention for Caregivers of Frail Older Chinese Adults: Testing an Intergenerational Caregiving Model
Brief Title: Mindfulness-Based Intervention for Caregivers of Frail Older Chinese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15604220
Record Dates: First submitted 2021-04-12; First posted 2021-04-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Frailty; Caregiver Burnout
MeSH Terms: conditions — Frailty; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief mindfulness based program (Experimental): A four session program, each last for 2.5 hours. Brief mindfulness exercises promote stress reduction, with an introduction of mindfulness to caregivers and home practice is encouraged with guidance.
  Interventions: Behavioral: Brief mindfulness based program
- Psychoeducation (Active Comparator): A four session program, each last for 2.5 hours. It promotes the coping and problem solving of caregivers. Brief home application included.
  Interventions: Behavioral: Psychoeducation
- Treatment-as-usual (No Intervention)

INTERVENTIONS:
Behavioral: Brief mindfulness based program — An intervention promotes the acceptance and emotion regulation in caregiving for frail older adults
  Arms: Brief mindfulness based program
Behavioral: Psychoeducation — An intervention promotes the coping and problem solving in caregiving for the frail older adults
  Arms: Psychoeducation

SUMMARY:
This is study to investigate the effects of a brief mindfulness-based program for frail older adults caregivers.

DETAILED DESCRIPTION:
The proposed study is a multi-site, three-arm randomized controlled trial of a mindfulness-based intervention for Chinese family caregivers in Hong Kong. Effects of the intervention will be compared with those of an evidence-based psychoeducation program, and treatment-as-usual. 240 caregivers of frail elderly with moderate to severe levels of frailty, will be recruited and randomly assigned to mindfulness-based intervention, psychoeducation, and treatment-as-usual experimental conditions. Overall program effectiveness will be analyzed on measures of caregiver burden, depression, anxiety, positive caregiving experience, spirituality, family conflict, and the biomarker of heart rate variability. Measures on coping styles, experiential avoidance, and self-efficacy will be explored to see if they mediate the changes to participant improvements in outcomes. 6-month follow-up will be included to investigate the maintenance effects.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of frail elderly based on a professional's assessment of Clinical Frailty Scale with a score of 6, indicating a moderate level of frailty or above (Rockwood et al., 2005)
* Caregivers being adult children or children in-law of the elder care receiver
* Caregivers who are experiencing caregiver burden at the time of study, with scores of 8 or above in Zarit Burden Interview-4

Exclusion Criteria:

* impairment, which may present difficulties in comprehending the content of the program
* Spouses, siblings, or friends will be excluded
* Caregivers of elders with moderate to severe dementia will be excluded and the Clinical Dementia Rating Scale will be administered
* Caregivers who had participated in an eight week Mindfulness-Based Stress Reduction or equivalent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Depression | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up
  assessed by a self-reported measure The Center for Epidemiologic Studies Depression Scale, 10 items, sum of scores from 0 to 30, the higher the score, the more severe in the depression symptoms

SECONDARY OUTCOMES:
Caregiver burden | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up.
  assessed by a self-reported measure Zarit Burden Interview, 22 items, sum of scores from 0 to 88, the higher the score, the more severe in the caregiver burden
Anxiety | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up
  assessed by a self-reported measure Hospital Anxiety and Depression Scale -Anxiety subscale, 7 items, sum of scores from 0 to 21, the higher the score, the more severe in the anxiety symptoms
Spiritual well-being | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up.
  assessed by a self-reported measure Functional Assessment of Chronic Illness, 12 items, sum of scores from 0 to 48, the higher the score, the better the level in well-being Therapy-Spiritual Well-Being Scale
family conflicts | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up
  assessed by a self-reported measure Revised Conflict Tactics Scale, 10 items, sum of scores from 0 to 40, the higher the score, the more severe in the level of family conflicts
Heart rate variability | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up.
  measured by the CorSense Heart Rate Variability monitor, the higher the heart rate variability, the better the ability to self-regulate in response to stressful situations
Coping styles | Change from pre-intervention, to 1-month follow-up, and to 6-month follow-up
  measured by a self-reported scale brief COPE, 28 items, sum of scores from 28 to 112, the higher the score, the better the level of positive coping

CONTACTS AND LOCATIONS:
Overall Officials: Herman, Hay-ming LO, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT04861610/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT04861610/ICF_001.pdf